CLINICAL TRIAL: NCT04988750
Title: An Open Label, Prospective, Pilot Study to Evaluate the Safety and Preliminary Efficacy of the Combination of Focused Ultrasound With Re-irradiation for the Treatment Patients With Recurrent Glioblastoma Multiforme Using NaviFUS System
Brief Title: Evaluate the Safety and Preliminary Efficacy of the Combination of NaviFUS System With Re-irradiation for rGBM Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NaviFUS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NF-2020-01
Record Dates: First submitted 2021-07-02; First posted 2021-08-03 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FUS + re-RT or FUS + SRS (Experimental): The SRS treatment will be administered for 3 consecutive days (one fraction of 7-9 Gy per day; total dose 21-27 Gy), including SRS treatment 1 (SRS 1), SRS treatment 2 (SRS 2), and SRS treatment 3 (SRS 3). At the SRS 1 and SRS 3, the patients will be shaved their hair at first, and the patient registration will be performed for the neuronavigation system according to the instruction of the system.
  cRT will be administered for 5 consecutive days within one week, and a full course is two weeks (one fraction of 3-4 Gy per day; total dose: 30-40 Gy), including cRT treatment 1 to cRT treatment 10 (cRT 1-cRT 10). At the cRT 1, cRT 3, cRT 6, and cRT 8, the patients will be shaved their hair at first, and the patient registration will be performed for the neuronavigation system according to the instruction of the system.
  Interventions: Device: NaviFUS System

INTERVENTIONS:
Device: NaviFUS System — Using the neuronavigator to precisely guide the ultrasound energy to brain tissues in real-time and intraoperatively.

SUMMARY:
This is an open label, single arm, prospective, and pilot study. Eligible patients will be enrolled after acquiring the signed informed consent and then will receive the treatment of re-RT combined with FUS (FUS + re-RT) on an outpatient basis. The re-RT in FUS + re-RT treatment will include fractioned stereotactic radiosurgery (SRS) treatment (FUS + SRS) or conventional radiotherapy (cRT) treatment (FUS + cRT). The treatment of SRS or cRT treatment given to patients is determined by the investigator depending on the volume and location of the treatment region.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male/female patients ≥ 20 years of age
2. Histologically proven glioblastoma multiforme (GBM) that is recurrent following standard radiation therapy (RT) and temozolomide and the second recurrent after prior treatment with an inhibitor of vascular endothelial growth factor (VEGF) or VEGFR (including bevacizumab) administration (bevacizumab failure).
3. Patients if already on the steroids then should be on a stable or decreasing dose of steroids for at least 7 days prior to study treatment
4. Minimum interval since completion of radiation treatment is 12 weeks.
5. At the time of study treatment, minimum interval since last drug therapy:

(1) 1 week for non-cytotoxic agents (e.g., interferon, tamoxifen), daily chemotherapy (e.g., metronomic temozolomide, cytoxan) or targeted therapies administered daily (e.g., gleevec, tarceva)

(2) 4 weeks since last cytotoxic therapy or inhibitor of VEGF or VEGFR (e.g., bevacizumab)

(3) 6 weeks since the completion of a nitrosourea-containing chemotherapy regimen (e.g., carmustine [BCNU])

6. Body mass index (BMI) ≥17 kg/ m2

7. Eastern Cooperative Oncology Group (ECOG) score ≤ 3

8. Patients with life expectancy ≥ 12 weeks

9. Adequate hepatic, renal, coagulation, and hematopoietic function.

1. Hemoglobin ≥ 8 g/dL
2. Platelets ≥ 100,000/mm3
3. Neutrophils ≥ 1,500/mm3
4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
5. Alanine transaminase (ALT) < 3 x ULN
6. Aspartate transaminase (AST) < 3 x ULN
7. Prothrombin time ≤ 1.2 x ULN
8. International Normalized Ratio (INR) < 1.5
9. Bilirubin < 2 x ULN

10. Patients with the region of interest (ROI) for FUS exposure are located at least 30 mm distance beneath the skull bone and the ROI is not in the deep center brain with crucial brain functions, such as in the region of brain stem, or motor or speech regions

11. Patients with the potential for pregnancy and their partner must agree to follow acceptable birth control methods to avoid conception. Female patients of child-bearing potential must have a negative pregnancy test.

12. Able to give written informed consent for the participation in the trial and comply with study requirements in the opinion of the investigator

Exclusion Criteria:

1. Patients with implanted pacemaker, defibrillator or deep brain stimulator, other implanted electronic devices in the brain or documented clinically significant arrhythmias
2. Patients with meningeal metastasis, intracranial stroke, congestive heart failure, unstable angina, cardiac arrhythmia, unstable cardiac status, and uncontrolled seizure activity
3. Patients with known HIV, however, that HIV testing is not required for entry into this study
4. Any patient requiring supplemental oxygen therapy
5. Use of any recreational drugs or history of drug addiction
6. Pregnant or breast-feeding women
7. The receipt of an investigational drug within a period of 28 days prior to the first FUS exposure
8. Known sensitivity/allergy to PET tracers, O-(2- [18F]fluoroethyl)- L-tyrosine (FET); Magnetic Resonance Imaging (MRI) contrast agents, Dotarem; Computer Tomography (CT) contrast agents; SonoVue®; or any of its components
9. Any other condition that, in the investigator's judgment, might increase the risk to the patients or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study
10. Abnormal baseline findings considered by the investigator to indicate conditions that might affect study endpoints
11. Patients who have acute hemorrhage within the ROI
12. Major surgery or significant traumatic injury that has not been recovered from by 4 weeks prior to screening, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤ 1 week prior to screening, or who have not recovered from side effects of such procedure or injury
13. Patients who have coagulopathy or risk factors for bleeding.
14. Receiving anticoagulants or antiplatelet drugs within one week before study entry
15. Receiving medications known to increase the risk of bleeding within one month before study entry (e.g., bevacizumab)
16. Contraindications to MRI, including but not limited to metallic implants and claustrophobia
17. Patients with severe hypertension (defined as systolic blood pressure > 180 mmHg or diastolic blood pressure >100 mmHg)
18. Patients with cardiac shunt
19. Patients with anticancer therapy-related adverse events which are unrecovered/unresolved to baseline or at grade 1 in severity

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 6 months
  Safety

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 6 months
  ORR based on Response Assessment in Neuro-Oncology (RANO) criteria
Progression-free survival (PFS) | Up to 6 months
  PFS and median PFS based on RANO criteria
Overall survival (OS) | Up to 6 months
  OS and median OS
Corticosteroid consumption | Up to 6 months
  Compared the steroid dosage before treatment and after treatment
Quality of life (QoL) | Up to 6 months

OTHER OUTCOMES:
Positron emission tomography (PET) uptake | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Medical Foundation, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No